CLINICAL TRIAL: NCT06773533
Title: Establishment of a Registry of Adjuvant Hormone-blockade Breast Cancer Patients Evaluated for Bone Mineral Metabolism
Brief Title: Registry of Adjuvant Hormone-blockade Breast Cancer Patients Evaluated for Bone Mineral Metabolism
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Als-BONE
Record Dates: First submitted 2024-12-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Establishment of a registry by which to census all patients treated with adjuvant hormone blockade for previous breast cancer in order to evaluate in future studies the trend of bone mass and its relationship to laboratoristic indices inherent in calcium metabolism, and the prevalence and incidence of fractures.

DETAILED DESCRIPTION:
Establishment of a registry by which to census all patients treated with adjuvant hormone blockade for previous breast cancer in order to evaluate in future studies the trend of bone mass and its relationship to laboratoristic indices inherent in calcium metabolism, and the prevalence and incidence of fractures.

Inclusion in the registry will be proposed consecutively to every patient with adjuvant hormone-blockade breast cancer diagnosed and evaluated at the Endocrinology Operative Unit for Bone Mineral Metabolism as part of the 'Diagnostic Clinical-Assistance Pathway (PDTA) of the patient with breast cancer' of IRCCS AOU of Bologna and referred/referred by Zamagni Oncology. The registry will include patients seen from 01/01/2015 for a duration of 15 years. A maximum follow-up duration for each patient is expected to be 10 years with an end date of enrollment on 12/31/2029 and a registry update deadline on 12/31/2039.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient undergoing adjuvant hormone blockade therapy (aromatase inhibitors, GnRH analogs, tamoxifen) for breast cancer referred by UO Oncology Zamagni
* Performed densitometry at UO Radiology Lovato and performed hematochemical tests inherent to mineral metabolism
* Informed consent obtained

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each breast cancer patient on adjuvant hormone blockade diagnosed and evaluated at the Endocrinology Operative Unit for Bone Mineral Metabolism as part of the 'Diagnostic Clinical Care Pathway (PDTA) of the Breast Cancer Patient' of IRCCS AOU of Bologna and referred/referred by Zamagni Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of a Registry for Patients Treated with Adjuvant Hormone Blockade for Breast Cancer: Evaluation of Bone Mass, Calcium Metabolism Indices, and Fracture Incidence | through study completion, an average of 15 years
  Establishment of a registry by which to census all patients treated with adjuvant hormone blockade for previous breast cancer in order to evaluate in future studies the trend of bone mass and its relationship to laboratoristic indices inherent in calcium metabolism, and the prevalence and incidence of fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Pagotto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No